CLINICAL TRIAL: NCT00025025
Title: Colorectal Cancer Screening: Fecal Blood vs. DNA
Brief Title: Screening Tests in Detecting Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: NCCTG-MC9944; P30CA015083 (NIH); MAYO-MC9944; NCCTG-MC9944; NCI-P01-0185
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm I: Participants eat no red meat and take no nonsteroidal anti-inflammatory drugs (NSAIDs) and no vitamin C or multivitamins for 3 days prior to and during stool sample collection. Participants collect stool samples 3 different times and perform fecal occult blood (FOB) test smears from each stool. After each collection, participants ship the whole stool and FOB test smear to their participating center for blinded multitarget DNA-based assay panel (MTAP) testing.
  Within 2 months after stool sample collection, participants have their blood drawn for additional MTAP testing and undergo colonoscopy.
  Interventions: Other: sample testing
- Arm II: Participants take no vitamin C or multivitamins for 3 days before and during stool sample collection. Participants collect stool samples and FOB test smears and samples are tested as in arm I.
  Within 2 months after stool sample collection, participants have their blood drawn for additional MTAP testing and undergo colonoscopy.
  Interventions: Other: sample testing

INTERVENTIONS:
Other: sample testing

SUMMARY:
RATIONALE: Screening tests may help doctors detect cancer cells early and plan more effective treatment for colorectal cancer.

PURPOSE: Randomized screening trial to compare the effectiveness of fecal occult blood testing with that of DNA-based testing of stool and blood in identifying colorectal cancer.

DETAILED DESCRIPTION:
Primary objectives:

1. To compare the performance characteristics (sensitivity, specificity, predictive values) of the fecal MTAP and most widely-used fecal occult blood test (Hemoccult) for identification of screen-relevant colorectal neoplasia (curablestage cancer and advanced adenomas with high-grade dysplasia/carcinoma in situ or size ≥ 1.0 cm.)
2. To evaluate the necessity of formal pretest preparation for MTAP by comparing the specificity of both the MTAP and Hemoccult tests in subject groups randomized to pre-test preparation versus no pre-test preparation.

Secondary objectives:

1. To compare detection rates of colorectal neoplasia by the fecal MTAP alone with those by flexible sigmoidoscopy (distal 60 cm of colonoscopic examination to serve as surrogate) and by the combination of sigmoidoscopy plus Hemoccult.
2. To characterize and compare the pathological and molecular features of screen-relevant colorectal neoplasms detected and not detected by the fecal MTAP.
3. To explore the sensitivity and specificity of the MTAP applied to plasma for the detection of screen-relevant colorectal neoplasia.
4. To maintain a specimen bank comprising stools and blood (plasma) from all subjects and tissue from screen-relevant neoplasms.

OUTLINE: This is a randomized, multicenter study. Participants are stratified according to age (50-64 [closed to accrual as of 6/5/03] vs 65-80), gender (male vs female), and participating center. Participants are randomized to one of two screening arms.

* Arm I: Participants eat no red meat and take no nonsteroidal anti-inflammatory drugs (NSAIDs) and no vitamin C or multivitamins for 3 days prior to and during stool sample collection. Participants collect stool samples 3 different times and perform fecal occult blood (FOB) test smears from each stool. After each collection, participants ship the whole stool and FOB test smear to their participating center for blinded multitarget DNA-based assay panel (MTAP) testing.
* Arm II: Participants take no vitamin C or multivitamins for 3 days before and during stool sample collection. Participants collect stool samples and FOB test smears and samples are tested as in arm I.

Within 2 months after stool sample collection, participants have their blood drawn for additional MTAP testing and undergo colonoscopy.

PROJECTED ACCRUAL: A total of 4,000 participants (2,000 per arm) will be accrued for this study.

ELIGIBILITY:
Required Characteristics:

1. ≥ 65 and ≤ 80 years of age.
2. Females must be postmenopausal (absence of menstrual periods for at least one year; patients on regular hormone replacement therapy; surgical intervention).

Contraindications:

1. FOBT screening ≤1 year prior to randomization.
2. Structural colorectal evaluation (i.e. colonoscopy, colon x-ray, or sigmoidoscopy) ≤10 years prior to randomization.
3. Overt rectal bleeding (hematochezia or melena) ≤1 month prior to randomization.
4. Prior colorectal resection for any reason.
5. Inability to stop therapeutic doses of NSAIDs (prophylactic doses of aspirin (≤325 mg) allowed [121] and Cox2 inhibitors (i.e. Celebrex, Vioxx) allowed.)
6. Coagulopathy or inablitity to discontinue anticoagulants (discontinuation must be superviesed by a physician).
7. Aerodigestive cancer ≤5 years prior to randomization.
8. Contraindications to colonoscopy (e.g., serious cardiopulmonary disease).
9. High-risk conditions for colorectal cancer (familial adenomatous polyposis, hereditary nonpolyposis colorectal cancer syndrome, other hereditary cancer syndromes, prior colorectal cancer or adenoma, inflammatory bowel disease, and

   * 2 first-degree relatives with colorectal cancer).
10. Chemotherapy ≤ 3 months prior to registration.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 -80 years
Sampling Method: Non-Probability Sample
Enrollment: 4482 (Actual)
Dates: Start 2001-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Ahlquist, MD, Study Chair — Mayo Clinic
Locations (65):
- United States (65):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tuscon, Arizona
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota